CLINICAL TRIAL: NCT02260895
Title: Almond Effects on Glucose Intolerance Study (AEGIS)
Brief Title: Almond Effects on Glucose Intolerance Study
Acronym: AEGIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Investigator left the institution.
Sponsor: Memorial Hermann Health System (Other)
Responsible Party: Principal Investigator, Aryn Knight, AVP Research, Memorial Hermann Health System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MH-14-0667
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard 2-hour 75-gram oral glucose tolerance test
- Almond Pre-test snack (Experimental): 1/2 ounce (14 g) almond snack 30 minutes prior to a 2-hour 75-gram oral glucose tolerance test
  Interventions: Dietary Supplement: Almond pre-test snack

INTERVENTIONS:
Dietary Supplement: Almond pre-test snack — unsalted, dry-roasted almonds, 1/2 oz (14 g), ingested 30 minutes prior to the start of a two-hour oral glucose tolerance test
  Other Names: unsalted, dry-roasted almonds
  Arms: Almond Pre-test snack

SUMMARY:
Diabetes is a major cause of morbidity and mortality worldwide. Prevention of diabetes is an important goal. The progression from impaired glucose tolerance to diabetes is thought to be promoted by the toxic effects of hyperglycemia on pancreatic beta cells. One of the main defects causing postprandial hyperglycemia in individuals with impaired glucose tolerance is reduced first phase (immediate) insulin release. The investigators hypothesis is that consuming a nutritional preload--a low-calorie, nutritionally balanced snack--30 minutes before ingesting a carbohydrate load, will moderate the hyperglycemic response to subsequent carbohydrate challenge and reduce glucotoxicity by stimulating insulin release and synthesis.

The aim of this study is to test this hypothesis by comparing the standard 75-gram, two-hour oral glucose tolerance test (OGTT) response of 30 fasting adults who have impaired glucose tolerance to their OGTT response when the test is preceded by ½ ounce (14 grams) of dry-roasted, unsalted almonds. A pre-load interval of 30 minutes was chosen so that the peak of phase 2 (delayed) insulin response to the pre-load (45-60 minutes) would coincide with the timeframe of the steepest OGTT rise in glucose (15 to 30 minutes post challenge).

The investigators hypothesize that the one-hour OGTT glucose level will be approximately 40 mg/dl lower when participants consume the pre-OGTT almond snack, compared to their one-hour glucose level on the standard two-hour OGTT. The two-hour OGTT glucose level is unlikely to show a statistically significant difference between the almond pre-test snack and control standard OGTT conditions.

DETAILED DESCRIPTION:
The study will be conducted at Physicians at Sugar Creek (PSC)-the model family practice center for the Memorial Family Medicine Residency Program. The ethnicity of PSC patients is approximately 30% non-Hispanic white, 30% Hispanic, 30% African-American, and 10% Asian.

Potential participants will be identified by searching PSC electronic medical records (Centricity) to find adults aged 18-75 with impaired glucose tolerance, without diabetes (one-hour oral glucose tolerance test result >160 md/dl and two-hour OGTT result <200 mg/dl), without hypoglycemic medications and corticosteroids on their active medications list, and without almond allergy on their allergy list.

Recruitment flyers will be posted in the clinic to encourage interested individuals to contact the investigators about their potential study eligibility. The investigators will also approach previously identified potentially eligible patients during routine clinical visits in the clinic, to elicit their interest in participating in the study. Those expressing interest will be scheduled for an intake visit with an investigator, to further ascertain their eligibility and invite eligible individuals to take part in the study. Interested eligible individuals who render verbal and written informed consent will then be instructed in the study protocol and scheduled for their first data gathering visit.

Each participant will be scheduled to undergo two 2-hour oral glucose tolerance tests (OGTT), starting between 7:00 and 9:30 a.m., one to four weeks apart. Test A will be a standard 75-gram OGTT. Test B will be an OGTT that will begin 30 minutes after ingestion of a low-carbohydrate pre-load "snack" consisting of 1/2 oz (14 grams) of unsalted, dry-roasted almonds (12 average size almonds). Each participant will be given an 8-ounce glass of water to drink with the almonds. Participants will be randomized to one of two test sequences (A-B or B-A), to control for sequence effects on results.

To minimize variability of OGTT results, participants will be asked to eat as they usually do throughout the study. Participants will be asked to refrain from vigorous physical activity for 8 hours prior to each OGTT and to minimize their physical activity during each OGTT. Participants will complete a Perceived Stress Scale and a 24-hour food, alcohol, and activity recall for the day before each OGTT to analyze potential confounding effects of stress, diet, alcohol, and physical activity on the results.

Blood sampling will be done for serial measurements of plasma glucose at time-zero, and at 60-minute intervals for two hours after each 75-gram glucose load. An investigator will monitor the timing of each blood draw closely to ensure timeliness. Blood will be drawn by one of two phlebotomists in the on-site laboratory and sent to the Memorial Hermann Southwest Hospital or Quest Lab (the latter only for the control OGTT, for patients whose insurance requires this) for analysis. The glucose results will be reported electronically to the patient's medical record in the routine manner for blood test results.

Investigators will abstract the glucose results from the patients' electronic medical records for data analysis purposes. The primary dependent variable is the mean difference in plasma glucose (fasting to 1-hr post 75-g glucose challenge, with vs. without snack. The secondary dependent variable is the mean difference in plasma glucose (fasting to 2-hr post 75-g glucose challenge, with vs. without snack). Student's t test will be used to analyze the differences between the standard 75-g OGTT results and the OGTT results following the almond pre-test snack. Analysis of variance will be used to analyze the data for confounding effects of ethnicity, gender, body mass index (BMI), and pre-test food and alcohol intake, physical activity, and perceived stress level.

Patients will receive their individual results and an investigator-generated evaluative commentary in a routine "lab letter". The results letter will be forwarded to each patient's primary care provider for review and appropriate clinical follow-up. Patients' results will be communicated scientifically in an aggregate manner, with no individual identifying information, to maintain patient confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* History of abnormal 1-hour OGTT result (>160 mg/dL) or 2-hour OGTT (>140)

Exclusion Criteria:

* History of a diagnosis of diabetes
* History of a 2-hour OGTT result >200 mg/dL
* History of a fasting glucose >125 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
One-hour OGTT result | 60 minutes into 2-hour oral glucose tolerance test
  One-hour oral glucose tolerance test result

SECONDARY OUTCOMES:
Two-hour OGTT result | 120 minutes into 2-hour oral glucose tolerance test
  Two-hour oral glucose tolerance test result (at 2 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Crouch, MD, MSPH, Principal Investigator — Memorial Hermann Health System
Locations (1):
- Physicians at Sugar Creek - Memorial Family Medicine Residency Program, Sugar Land, Texas, United States